CLINICAL TRIAL: NCT04954755
Title: Development and Validation of a Prediction Model for Refeeding Syndrome in ICU Patients Undergoing Enteral Nutrition
Brief Title: Development and Validation of a Prediction Model for Refeeding Syndrome in ICU Patients Undergoing Enteral Nutrition Patients
Acronym: RFS
Status: Completed | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-394
Record Dates: First submitted 2021-07-06; First posted 2021-07-08 (Actual); Last update posted 2021-07-08 (Actual); Status verified 2021-06

CONDITIONS: Development and Validation of a Prediction Model for Refeeding Syndrome in ICU Patients Undergoing Enteral Nutrition
Keywords: Refeeding Syndrome;Enteral Nutrition;Prediction;Intensive Care

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- RFS
- non-RFS

SUMMARY:
This study intends to strengthen the discussion on the risk factors of RFS in critically ill patients, and construct an RFS risk prediction model which is easy for clinical medical staff to use and has a high sensitivity and specificity; In order to help medical staff to identify the high-risk groups of RFS in critically ill patients efficiently and accurately, and take targeted care and treatment for patients, so as to reduce the adverse consequences of RFS on critically ill patients.

ELIGIBILITY:
Inclusion Criteria:

* (1) Age ≥18 years old; (2) Patients with mechanical ventilation; (3) First admission to ICU； (4) The time of receiving enteral nutrition support in ICU was ≥ 3 days.

Exclusion Criteria:

* (1)Ppregnant women or lactating patients;(2) Patients with incomplete information;(3) There are other risk factors leading to hypophosphatemia, such as continuous hemodialysis , hyperphosphatemia treatment,Parathyroid gland resection was performed within 3 months.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Modeling queue: Relevant information of 433 patients who received enteral nutrition from January 2018 to July 2020 in ICU of a tertiary hospital in Zhejiang .
  Authentication queue: Relevant information of 120 patients who received enteral nutrition from August 2020 to October 2020 in ICU of four tertiary hospitals in Zhejiang .
Sampling Method: Non-Probability Sample
Enrollment: 553 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2020-10-31 (Actual); Study Completion 2020-10-31 (Actual)

PRIMARY OUTCOMES:
Occurrence of RFS | from December 1, 2019 to October 31, 2020
  Occurrence of RFS：Within 72 hours after feeding serum phosphorus < 0.0.87mmol/L, or from the baseline levels drop > 0.16% or drop > 30%;And (or) hypokalemia, hypomagnesemia, hypocalcemia and corresponding clinical symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Meiqi Yao, undergraduate, Study Chair — Second Affiliated Hospital, School of Medicine, Zhejiang University; Xingxia Long, postgraduate, Principal Investigator — Huzhou University
Locations (1):
- Development and Validation of a Prediction Model for Refeeding Syndrome in ICU Patients Undergoing Enteral Nutrition, Hanzhou, Zhejiang, China